CLINICAL TRIAL: NCT07090551
Title: Effect of Occlusal Splint on Head and Neck Muscles in Patients With Bruxism and Myofascial Pain: An Ultrasonographic Study
Brief Title: Effect of Occlusal Splint on Head and Neck Muscles in Patients With Bruxism and Myofascial Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Berk Bilgen, research assistant, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/130
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Myofacial Pain Syndrome; Local Myalgia; Masticatory Muscle Pain; Bruxism
Keywords: myofacial pain syndrome; bruxism; ultrasonography; occlusal splint; masseter muscle; splenius capitis muscle
MeSH Terms: conditions — Facial Neuralgia; Bruxism

STUDY DESIGN:
Intervention Model Description: Patients who present with various temporomandibular disorder (TMD) complaints to the "Temporomandibular Disorders Clinic" of the Department of Prosthodontics at Istanbul University Faculty of Dentistry undergo routine clinical examinations, during which TMD-DC (Diagnostic Criteria for Temporomandibular Disorders) forms are completed to aid in reaching an accurate diagnosis. Based on clinical findings and form results, patients suspected of having masticatory muscle disorders but lacking a definitive diagnosis are referred for ultrasonographic (USG) imaging to investigate potential myofascial trigger points, pathological changes, or muscle atrophy in the masticatory muscles.
  Subsequently, USG results are evaluated in conjunction with the clinical findings and TMD-DC assessments to establish a definitive diagnosis. If the presence of myospasm or myofascial pain syndrome originating from the masseter and/or temporalis muscles is confirmed, occlusal splint therapy is init
Who Masked: Outcomes Assessor
Masking Description: The researcher performing the ultrasonographic imaging is blinded to the group allocation of the patients. The study is designed as a single-blind trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Patients in the control group present with myofascial pain; however, no treatment will be administered to them. Ultrasonographic images taken at baseline and at the end of the three-month period will be compared both within the control group and with the patient group receiving occlusal splint therapy.
- occlusal splint group (Experimental): Ultrasonographic imaging will be performed on patients with myofascial pain who undergo occlusal splint therapy, both prior to treatment and at the end of the treatment period (three months after the initiation of therapy). These data will be compared within the treatment group and against the control group.
  Interventions: Device: occlusal splint therapy

INTERVENTIONS:
Device: occlusal splint therapy — Patients with myofascial pain will receive occlusal splint therapy, which is a clinically accepted treatment method.
  Arms: occlusal splint group

SUMMARY:
The study group will be selected from patients who previously presented with various temporomandibular disorder (TMD) complaints to the "Temporomandibular Disorders Clinic" of the Department of Complete and Removable Dentures at the Faculty of Dentistry, Istanbul University. During routine examinations, TMD-DC (Diagnostic Criteria for Temporomandibular Disorders) forms are completed to aid in achieving an accurate diagnosis. Subsequently, patients suspected of having TMD of masticatory muscle origin but without a definitive diagnosis are routinely referred for ultrasonographic (USG) imaging. Patients meeting these criteria will be included in the study.

Participants will be divided into two groups. The first group will consist of patients who have already undergone USG imaging during their routine examination, have been definitively diagnosed with masticatory muscle disorders based on clinical and radiographic findings, and have initiated routine occlusal splint therapy in the clinic. The 12-week treatment process of these patients will not be altered in any way. At the final follow-up session after the 12-week routine treatment protocol, the TMD-DC form completed at baseline will be re-administered, and the two forms will be compared to evaluate changes in symptoms and pain levels. Another USG imaging will also be performed at this session.

The second group, serving as the control group, will include patients who have previously undergone USG imaging during routine examination and have received a definitive diagnosis of masticatory muscle disorders based on clinical and radiographic evaluations, but have not yet begun treatment. Patients whose turn for treatment begins during the study period will be excluded from this group. At the end of the 12-week period, the TMD-DC form will be re-administered, and a second USG imaging will be performed. This process will not interfere with the patients' position in the treatment queue, and treatment will commence as scheduled. In the second USG session, changes in the thickness and elasticity of the masseter, temporalis, trapezius, sternocleidomastoid, and splenius capitis muscles will be assessed by comparing the two imaging records.

DETAILED DESCRIPTION:
The study is designed as a prospective observational clinical research. The study group will consist of patients who previously presented with various temporomandibular disorder (TMD) complaints to the "Temporomandibular Disorders Clinic" of the Department of Prosthodontics at the Faculty of Dentistry, Istanbul University. During routine examinations, patients are asked to complete the TMD-DC (Diagnostic Criteria for Temporomandibular Disorders) forms to facilitate accurate diagnosis. Subsequently, patients who are suspected of having TMD of masticatory muscle origin but for whom a definitive diagnosis cannot be established are routinely referred for ultrasonographic (USG) imaging. Patients who meet these criteria will be included in the study.

Participants will be divided into two groups. The first group will comprise patients who have previously undergone USG imaging for routine diagnostic purposes, have been definitively diagnosed with masticatory muscle disorders based on clinical and radiographic examinations, and have initiated occlusal splint therapy as part of routine clinical care. The 12-week treatment protocol of these patients will not be altered in any way. At the final follow-up session at the end of the 12-week treatment period, the TMD-DC form previously completed at baseline will be re-administered, and the two forms will be compared to evaluate changes in patients' symptoms and pain levels. Additionally, a second USG imaging will be performed at this session.

The second group will consist of patients who have undergone USG imaging for routine diagnostic purposes, have been definitively diagnosed with masticatory muscle disorders based on clinical and radiographic findings, but have not yet begun treatment due to waiting their turn in the treatment queue. Patients who start occlusal splint therapy during the study period will be excluded from the control group. This group will serve as the control group of the study. At the end of the 12-week observation period, participants in this group will again complete the TMD-DC form and undergo a second USG imaging. This process will not affect their place in the treatment queue, and treatment will be initiated when their turn arrives.

In the final USG session, the thickness and elasticity of the masseter, temporalis, trapezius, sternocleidomastoid, and splenius capitis muscles will be compared between the two imaging sessions. In this way, the effects of occlusal splints on the morphology and elasticity of the head and neck muscles will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients who have presented to the Faculty of Dentistry at Istanbul University with temporomandibular disorder (TMD) complaints, Patients diagnosed with myospasm and/or myofascial pain syndrome in the masseter and/or temporalis muscles prior to treatment, Patients with no physical or mental disabilities, Patients over the age of 18, Patients who have not previously received any treatment for TMD.

Exclusion Criteria:

Patients with any type of TMD other than masticatory muscle disorders, Patients who have previously received any form of TMD treatment, Patients under the age of 18.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
ultrasonography results | 3 months
  The masseter, temporalis, sternocleidomastoid, splenius capitis, and trapezius muscles will be evaluated using ultrasonography. For each muscle, elastography values, thickness at rest, and thickness during maximum clenching will be measured. All parameters will be recorded both before the initiation of treatment and three months after treatment, and the values will be compared accordingly.

SECONDARY OUTCOMES:
dc/tmd form results | 3 mouths
  Through the use of DC/TMD forms, all patients in both groups will undergo assessments of mandibular movements, muscle palpation findings, the degree of functional jaw limitation, depression and anxiety questionnaires, and pain questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: berk bilgen, phd, Principal Investigator — Istanbul University; olcay şakar, phd, prof., Study Director — Istanbul University
Locations (1):
- Istanbul University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yalcin ED, Aslan Ozturk EM. Ultrasonographic evaluation of the effect of splint therapy on masseter muscle and blood flow in patients with bruxism. Cranio. 2025 Jan;43(1):135-143. doi: 10.1080/08869634.2022.2088575. Epub 2022 Jul 11. PMID 35816105
- [Background] Bilgen B, Akpinar E, Tepe RD, Karabas HC, Sakar O. Effects of occlusal splint therapy on the masseter and temporalis muscles in female patients with myofascial pain syndrome: An ultrasonographic study. Cranio. 2025 Sep;43(5):868-878. doi: 10.1080/08869634.2025.2490297. Epub 2025 Apr 22. PMID 40264294